CLINICAL TRIAL: NCT05072366
Title: Reliability and Validity of the Turkish Version of the Tinetti Fall Efficacy Scale in Older People and Comparison With Other Fall Scales
Brief Title: Reliability and Validity of the Turkish Version of the Tinetti Fall Efficacy Scale in Older People
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Melahat Selin DURMUŞ, Physiotherapist, Kırıkkale University
Other Study IDs: KırıkkaleUniversityMSD
Record Dates: First submitted 2021-09-19; First posted 2021-10-08 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Fall Patients
Keywords: Falling; Gait; Balance; Geriatrics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Joint International Commission (JCI) defines a fall as an unplanned, abrupt, change of motion towards the ground that may result in physical injury. Falls are among the most obvious reasons for applying to health centers after an involuntary external injury. Risk of falls diagnostic tools; It is used to reduce the incidence of falls, to reduce the severity of falls, to increase walking and existing functional status, to determine the factors causing falls and to keep them under control, and to raise awareness of health personnel about falls. This study aims to make the Turkish cultural adaptation of the Tinetti Fall Efficiency Scale, to test the validity and reliability of the factorial structure in elderly individuals. It was planned to determine that it is specific and sensitive. The Fall Efficiency Scale (DAS) was developed based on the definition of this fear as "low perceived self-efficacy in avoiding falls during harmless activities of daily living".

DETAILED DESCRIPTION:
Is the fall effectiveness scale an effective scale that determines the fear of falling? To find the answer to this question of which scale is more sensitive when compared to other scales, to ensure the adaptation of the elderly individuals in Turkish society and to raise awareness of the discomforts that can be experienced after falling to the geriatric individual and their surroundings, as a result of this, by enabling those at risk of falling to contact health professionals, preventive rehabilitation and other treatment methods are encouraged. It is aimed to gain public awareness about reducing health expenditures and protecting body integrity.

This thesis study is suitable for the methodological research method that investigates the validity and reliability of a questionnaire. In this study demographic data (age, gender, educational status, occupation, marital status) of individuals will be questioned in the initial evaluations. Height (m), weight (kg) will be recorded and body mass index (BMI) will be determined as body weight/height2 (kg/m2). The drugs used, co-morbidities, backgrounds will be recorded in the socio-demographic information forms of the individuals will be applied. This study aimed to adapt the Tinetti Fall Effectiveness Scale (FES), a tool to measure fear of falling, into Turkish, to demonstrate its validity-reliability and sensitivity to change in elderly individuals, and to compare the Timed Up and Go Test, Fall Risk Self-Assessment Scale, Tinetti Balance, and Gait Assessment and Activity. Together with the Specific Balance Confidence scales, an answer was sought for the question of which is the most effective scale for falling.

In scale studies, taking at least 3 or 5-10 people for each scale item constitutes the sample size. As the Fall Efficiency Scale consisted of 10 items, it was planned to study with 51 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years old and over,
* Not having a cooperation problem (individuals with a mini mental test score >24),
* Not having communication difficulties or problems
* Voluntarily accepts participation in the research.

Exclusion Criteria:

* Those with uncontrollable hypertension, heart disease, cardiac arrhythmia, cardiovascular disease,
* Those who have malignancy and cause malignancy, receive chemotherapy, radiotherapy,
* Those who have any neurological or orthopedic disorder that will disrupt the balance,
* Individuals who are addicted to alcohol and drugs,
* Those who do not accept to participate in the research.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: It is planned to conduct a study with elderly inpatients at the Izmir Governor's Private Empathy Care Center.
  Turkish volunteers aged 65 and over.
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Socio-demographic Information Form | through study completion, an average of six months
  Demographic data of individuals (age, gender, educational status, occupation, marital status) will be questioned. Height (m), weight (kg) were recorded and body mass index (BMI) will be determined as body weight/height2 (kg/m2). Medications used, additional diseases, backgrounds will be recorded in the socio-demographic information forms of the individuals.
Standardized Mini Mental Test | through study completion, an average of six months
  The scale, which consists of 11 items, gathered under five main headings as orientation, recording memory, attention and calculation, recall and language, is evaluated over a total of 30 points. While the maximum score on this scale is 30, scores below 20 in adults indicate cognitive impairment. The ideal threshold value of MMDT was found to be 24.
Fall Efficacy Scale | through study completion, an average of six months
  Evaluates the activities of daily living in 10 different activities by scoring "on a scale of 1 to 10, where 1 is very confident and 10 is very confident, how sure are you that you can do the following activities without falling?"; A total score above 70 indicates that the person has a fear of falling.
Fall Risk Self-Assessment Scale | through study completion, an average of six months
  It is a scale that evaluates the risk of falling in the elderly. It consists of 13 items assessing the risk of falling in the elderly. The answers are yes (1 point) and no (0 points), and individuals who score 4 points or more from the score are classified as having a high risk of falling.
Activity-Specific Balance Confidence Scale | through study completion, an average of six months
  Individuals were asked 16 questions about how confidently they performed the movements they performed during daily life and were asked to give a score between 0 and 100.
  At the end of the test, the scores were summed up and divided by 16 to obtain the individual's ABC score. A high value indicates that the individual feels confident about balance.
Time up and go | through study completion, an average of six months
  A score ≥ 13.5 s indicated a high risk of falling. The patient was asked to get up from the chair he was sitting in, walk 3 meters (at his own walking pace), then go back and sit on the chair again, and the total time spent was recorded. The patient was allowed to use the arm of the chair when getting up from the chair and to use an assistive device during this test.
Tinetti Balance and Gait Test | through study completion, an average of six months
  In the test used to evaluate balance, the walking score is a maximum of 12 points, the balance score is a maximum of 16 points and a total of 28 points. Those who score twenty-six and below are considered to have a problem. Studies have shown that the lower the score, the higher the risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Melahat S. DURMUŞ, PT, Study Chair — Kırıkkale University; Meral SERTEL, Assoc. Prof, Study Director — Kırıkkale University; Saniye AYDOĞAN, Dr., Study Director — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The main test of the thesis to be valid and reliable — https://instruct.uwo.ca/kinesiology/9641/Assessments/Biological/FES.html